CLINICAL TRIAL: NCT00950027
Title: Prospective Randomized Double Blind Study Comparing the Effect of Oropharyngeal Decontamination by Povidone-iodine to Placebo on Ventilator-associated Pneumonia in Patients With Head Trauma or Cerebral Hemorrhage
Brief Title: Study of Povidone Iodine to Reduce Pulmonary Infection in Head Trauma and Cerebral Hemorrhage in Intensive Care Unit
Acronym: SPIRIT-ICU
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: Rennes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: EudraCT 2006-006353-27; AFSSAPS A70642-35 (Other: AFSSAPS: French Health Products Safety Agency); Sponsor PHRC/06-05 SPIRIT ICU (Other: Rennes University Hospital)
Record Dates: First submitted 2009-07-30; First posted 2009-07-31 (Estimated); Last update posted 2012-07-06 (Estimated); Status verified 2012-07

CONDITIONS: Ventilator Associated Pneumonia
MeSH Terms: conditions — Pneumonia, Ventilator-Associated | interventions — Povidone-Iodine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- povidone iodine (Experimental): Povidone iodine
  Interventions: Drug: povidone iodine
- placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: povidone iodine — oropharyngeal decontamination every 4 hours
  Arms: povidone iodine
Drug: Placebo — oropharyngeal decontamination every 4 hours
  Arms: placebo

SUMMARY:
Head trauma and severe cerebral hemorrhage are major risk factors for development of ventilator-associated pneumonia. In a previous open labelled, single center study the investigators showed that repeated oropharyngeal decontamination with povidone-iodine may be an effective strategy to decrease the prevalence of ventilator-associated pneumonia in patients with head trauma. The present study aims to confirm these results in a multicenter, double blind study including patients suffering from head trauma or cerebral hemorrhage.

ELIGIBILITY:
Inclusion Criteria:

* Adults > 18 years
* Closed head trauma with a Glasgow Coma Score <=8 or cerebral Hemorrhage with a Glasgow Coma Score of <=8
* Expected need mechanical ventilation for >=2 days
* Written informed consent from the patient's next-of-kin. If no relative is present at the time of inclusion, the patients will be included according to the emergency procedure

Exclusion Criteria:

* Impossibility to perform oropharyngeal decontamination within 12 h following the initial episode
* Facial injury with impossibility to perform the oropharyngeal decontamination
* Tetraplegia
* Known history of reaction to iodine
* Respiratory disease or pulmonary infiltrate(s) at inclusion
* Need for curative antibiotics
* Mercurial antiseptics treatment
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 179 (Actual)
Dates: Start 2008-04; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Rate of ventilator associated pneumonia | 30 days

SECONDARY OUTCOMES:
Time to ventilator associated pneumoniae | 30 days
Rate of early (<=7 days) and late (>7 days) ventilator associated pneumoniae | 30 days
Length of mechanical ventilation | 30 days
Other infections | 30 days
Acute respiratory distress syndrome | 30 days
Treatments administered (antibiotics, sedatives, transfusion) | 30 days
Length of ICU and hospital stay | Hospital discharge
Death | ICU, 1 months, 3 months
Oropharyngeal bacterial colonisation | 30 days
Type of anesthetic agents received | 30 days
Rate of tracheostomy | 30 days
Rate of transfusion (red blood cells, platelets, plasma) | 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Philippe Seguin, MD, PhD, Principal Investigator — Rennes University Hospital; Bruno Laviolle, MD, Study Chair — Rennes University Hospital
Locations (7):
- France (7):
  - CHU Angers, Angers
  - Réanimation chirurgical Hopital Hotel Dieu-CHU de Nantes, Nantes
  - CHU de Poitiers, Poitiers
  - Surgical Intensive Care Unit - CHU de Rennes, Rennes
  - CHU de Rouen, Rouen
  - Réanimation chirurgicale CHU Tours, Tours
  - CHG Vannes, Vannes

REFERENCES:
- [Derived] Seguin P, Laviolle B, Dahyot-Fizelier C, Dumont R, Veber B, Gergaud S, Asehnoune K, Mimoz O, Donnio PY, Bellissant E, Malledant Y; Study of Povidone Iodine to Reduce Pulmonary Infection in Head Trauma and Cerebral Hemorrhage Patients (SPIRIT) ICU Study Group; AtlanRea Group. Effect of oropharyngeal povidone-iodine preventive oral care on ventilator-associated pneumonia in severely brain-injured or cerebral hemorrhage patients: a multicenter, randomized controlled trial. Crit Care Med. 2014 Jan;42(1):1-8. doi: 10.1097/CCM.0b013e3182a2770f. PMID 24105456